CLINICAL TRIAL: NCT05428605
Title: In Vitro Study of the Efficacy of Different Immunomodulators on the Th17/Treg Balance in a Cohort of Relapsed Membranous Nephropathy
Brief Title: In Vitro Immunomodulation in Membranous Nephropathy Relapses
Acronym: BIOGEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-AOIP-06
Record Dates: First submitted 2022-06-10; First posted 2022-06-23 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Extramembranous Glomerulopathy
Keywords: membranous nephropathy; immunomodulation; relapse; Th17/Treg pathways
MeSH Terms: conditions — Glomerulonephritis, Membranous; Recurrence | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: To compare in vitro the effect of different immunomodulators on Th17/Treg lymphocyte balance in a cohort of relapsed MN patients to determine the best therapeutic approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GEM patients (Experimental)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — 10 mL on lithium heparinate tubes, 10 mL on EDTA tubes.

SUMMARY:
In order to propose the best therapeutic option to relapsed MN patients with strong activation of the Th17 pathway, the investigators propose to study in vitro the effect of different immunomodulators on the Th17/Treg balance, assessed by cytokine profile and lymphocyte phenotyping using flow cytometry.

DETAILED DESCRIPTION:
Membranous Nephropathy (MN) is a rare autoimmune renal disease and the first cause of nephrotic syndrome in adults. In one third of cases, it progresses to end-stage renal failure. Rituximab has shown very good efficacy (60-80%) and excellent safety in this indication. However, one third of MN patients relapse after a course of rituximab, raising the question of maintenance treatment or repeated courses of rituximab whose long-term impact is unknown.

The investigators studied the cytokine profile of MN patients and demonstrated, after non-specific stimulation of innate immunity cells and T cells, a Th17 profile (increased levels of interleukin-6 (Il-6) and interleukin-17A (Il-17A) compared to healthy subjects), and inhibition of the Th1 (decreased IL-12p70 and Interferon-γ (IFN-γ)) and T regulatory T reg pathways (decreased IL-10) (doi: 10. 3389/fimmu.2020.574997).

Th17 cells and Treg cells with interconnected development have opposite roles. Th17 cells induce inflammation to initiate a reaction against a pathogen, while Treg cells control an inflammatory reaction.

The investigators showed that high Il-17A levels were associated with a risk of thrombotic events (p = 0.03) and relapse (p = 0.0006). A patient with an IL-17A level > 73 pg/ml had a 10.5-fold increased risk of relapse.

Rituximab-induced remission leads to an increase in Treg and Th1 pathway cytokines but has no impact on IL-17A production, which remains important even in remission.

Thus, in this group of patients with high IL-17A levels, targeted action on B lymphocytes is probably not sufficient to avoid relapse and the addition of a treatment aimed at inhibiting the Th17 pathway and promoting Treg induction seems legitimate.

Various potential treatment exist: anti-Il-6 antibodies (tocilizumab), anti-Il-17 antibodies (secukinumab), low-dose Il-2 (a few studies have demonstrated its ability to induce Treg in various autoimmune diseases), hydroxychloroquine in low doses (used in lupus to limit relapses and having an anti-inflammatory effect), the plant extract Alphanosos (anti-Th1) or Levamizole (validated in nephrotic syndrome in children).

In order to propose the best therapeutic option to relapsed MN patients with a strong activation of the Th17 pathway, the investigators propose to study in vitro the effect of these different immunomodulators on the Th17/Treg balance evaluated by cytokine profile and lymphocyte phenotyping in flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patient with MN proven on renal biopsy or by the presence of anti-PLA2R1 or anti-THDS71 antibodies
3. Relapsed MN, defined as proteinuria > 3.5g/g after achieving remission (partial or complete, definitions according to KDIGO 2012 guidelines)
4. At a distance from any immunosuppressive treatment (at least 6 months)
5. Freely given informed consent signed by the patient after clear, fair and appropriate information
6. Affiliated to a social security system

Exclusion Criteria:

1. Pregnant or breastfeeding woman
2. Patient under 18 years of age
3. Persons of legal age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Cytokine ELISA profiles of the Th17 pathway (IL-17 level), the Treg pathway (IL-10 level), the Th1 pathway (IL-12p70, IFN-γ) and the Th2 pathway (IL-4 and IL-5) | 18 months
  All cytokines (IL-17, IL-10, IL-12p70, IFN-γ, IL-4 and IL-5) measured by ELISA will be expressed in pg/ml.

SECONDARY OUTCOMES:
Lymphocyte phenotyping (Treg and Th17) determined by flow cytometry | 18 months
  Percentage of cells expressing the fluorescent marker of interest

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No
IPD is not planned to be shared with other researchers than the investigators